CLINICAL TRIAL: NCT04268160
Title: Glutathione Peroxidase Activity in Subjects With Aortic Stenosis Undergoing Transcatheter Aortic Valve Replacement.
Brief Title: GPx Activity in Subjects With Aortic Stenosis Undergoing TAVR
Status: Withdrawn | Type: Observational
Why Stopped: Funding issues and closed with the IRB
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201902486
Record Dates: First submitted 2020-02-05; First posted 2020-02-13 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Glutathione Peroxidase Activity; Aortic Stenosis; Transcatheter Aortic Valve Replacement
Keywords: glutathione peroxidase, GPx, aortic stenosis, transcatheter aortic valve replacement, TAVR
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with severe aortic stenosis undergoing TAVR: GPx activity levels will be measured on the day of TAVR procedure, the day of discharge, 1 month, and 6 months after the procedure
  Interventions: Diagnostic Test: Blood draw to measure GPx activity; Diagnostic Test: Blood draw to measure SOD activity; Diagnostic Test: Blood draw to measure Lp(a) levels
- Patients without aortic stenosis: GPx activity levels will be measured on day of recruitment
  Interventions: Diagnostic Test: Blood draw to measure GPx activity; Diagnostic Test: Blood draw to measure SOD activity; Diagnostic Test: Blood draw to measure Lp(a) levels

INTERVENTIONS:
Diagnostic Test: Blood draw to measure GPx activity — Routine blood draw to measure levels of blood markers.
Diagnostic Test: Blood draw to measure SOD activity — Routine blood draw to measure levels of blood markers.
Diagnostic Test: Blood draw to measure Lp(a) levels — Routine blood draw to measure levels of blood markers.

SUMMARY:
The aim of this project is to investigate the association of glutathione peroxidase (GPx) and severe aortic stenosis (AS), as well as the impact of transcatheter aortic valve replacement (TAVR) on GPx activity post-procedure. The burden of oxidative stress will be determined by the measurement of GPx, superoxide dismutase (SOD) and lipoprotein A (Lp(a)). We hypothesize GPx activity is reduced in participants with severe AS vs control groups and GPx activity is to increase after TAVR is performed.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Patients with severe AS including participants with low flow, low gradient severe AS and paradoxical severe AS
* Patients meeting criteria for TAVR procedure

Exclusion Criteria:

* Previous aortic valve replacement (surgical or TAVR)
* Participants undergoing chemotherapy
* End stage liver disease/cirrhosis (liver produces GSH)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants with severe aortic stenosis undergoing TAVR. They will be matched with patients without aortic stenosis based on age, gender, race, and co-morbidities (including stroke, history of coronary artery disease, heart failure, diabetes, hypertension, and other valvular diseases).
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-11 (Estimated); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Level of GPx in blood samples | Baseline up to 6 months
  Glutathione peroxidase activity levels measured from whole blood in U/L units in participants with severe aortic stenosis after transcatheter valve replacement compared with the matched population

CONTACTS AND LOCATIONS:
Overall Officials: Chinelo Udemgba, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Redfors, B. A. (2017). Biomarkers in Aortic Stenosis: A systematic Review. Structural Heart. The Journal of the Heart Team, 1-13.
- [Background] Otto CM. Aortic stenosis and hyperlipidemia: establishing a cause-effect relationship. Am Heart J. 2004 May;147(5):761-3. doi: 10.1016/j.ahj.2003.12.014. No abstract available. PMID 15131528
- [Background] Memet C, Gerede DM, Ozenci M, Akbulut IM, Acibuca A, Kilickap M, Erol C. Evaluation of the Role of Oxidative Stress in Degenerative Aortic Stenosis. J Heart Valve Dis. 2015 Jul;24(4):445-50. PMID 26897814
- [Background] Nimse, S. B. (2015). Free radicals, natural antioxidants, and their reaction mechanism. Royal Society of Chemistry, 27986-28006.
- [Background] Blankenberg S, Rupprecht HJ, Bickel C, Torzewski M, Hafner G, Tiret L, Smieja M, Cambien F, Meyer J, Lackner KJ; AtheroGene Investigators. Glutathione peroxidase 1 activity and cardiovascular events in patients with coronary artery disease. N Engl J Med. 2003 Oct 23;349(17):1605-13. doi: 10.1056/NEJMoa030535. PMID 14573732
- [Background] Bolzan AD, Bianchi MS, Bianchi NO. Superoxide dismutase, catalase and glutathione peroxidase activities in human blood: influence of sex, age and cigarette smoking. Clin Biochem. 1997 Aug;30(6):449-54. doi: 10.1016/s0009-9120(97)00047-7. PMID 9316738
- [Background] Zheng KH, Tsimikas S, Pawade T, Kroon J, Jenkins WSA, Doris MK, White AC, Timmers NKLM, Hjortnaes J, Rogers MA, Aikawa E, Arsenault BJ, Witztum JL, Newby DE, Koschinsky ML, Fayad ZA, Stroes ESG, Boekholdt SM, Dweck MR. Lipoprotein(a) and Oxidized Phospholipids Promote Valve Calcification in Patients With Aortic Stenosis. J Am Coll Cardiol. 2019 May 7;73(17):2150-2162. doi: 10.1016/j.jacc.2019.01.070. PMID 31047003
- [Background] Arsenault BJ, Boekholdt SM, Dube MP, Rheaume E, Wareham NJ, Khaw KT, Sandhu MS, Tardif JC. Lipoprotein(a) levels, genotype, and incident aortic valve stenosis: a prospective Mendelian randomization study and replication in a case-control cohort. Circ Cardiovasc Genet. 2014 Jun;7(3):304-10. doi: 10.1161/CIRCGENETICS.113.000400. Epub 2014 Apr 5. PMID 24704946
- [Background] Mahmaljy H, Tawney A, Young M. Transcatheter Aortic Valve Replacement. 2023 Jul 24. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK431075/ PMID 28613729